CLINICAL TRIAL: NCT05252637
Title: Laparoscopic Fascial Duplication Plus Sacral Colpopexy in Posterior Vaginal Prolapse: a Randomized Clinical Trial
Brief Title: Laparoscopic Fascial Duplication Plus Sacral Colpopexy in Posterior Vaginal Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Principal Investigator, Andrea Morciano, Panico Pelvic Floor Center, Azienda Ospedaliera Cardinale G. Panico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1202TricaseLSC
Record Dates: First submitted 2022-02-13; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Pelvic Organ Prolapse; Posterior Vaginal Wall Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duplication plus LSC (Experimental): Laparoscopic duplication of posterior vagina plus mesh placement
  Interventions: Procedure: Laparoscopic Fascial Posterior Vagina Duplication
- LSC (No Intervention): Laparoscopic Sacral Colpopexy with mesh placement on posterior vagina

INTERVENTIONS:
Procedure: Laparoscopic Fascial Posterior Vagina Duplication — Laparoscopic Fascial Posterior Vagina Duplication with absorbable sutures for posterior prolapse (plus standard Sacral Colpopexy)
  Arms: Duplication plus LSC

SUMMARY:
A Randomized Clinical Trial on Laparoscopic Fascial posterior vaginal duplication with absorbable sutures plus sacral colpopexy mesh placement VS sacral colpopexy isolated for vaginal posterior prolapse

DETAILED DESCRIPTION:
Laparoscopic sacral colpopexy is the gold standard procedure for pelvic organ prolapse. Anyway, vaginal fascial surgery is already considered the most appropriate for posterior vaginal prolapse. This prospective randomized pilot study is aimed to verify if the combination of laparoscopic duplication of vaginal fascia with absorbable sutures could increase benefits of sacral colpopexy on the posterior vagina in terms of prolapse (evaluating 1 year POP-Q).

Secondary endpoints of this comparison are incidence of intra- or postoperative complications estimated blood loss, postoperative pain (evaluated by VAS), days of hospitalization and costs for the health care system.

Statistical Analysis and Study Design This is a single Institution prospective randomized clinical trial conducted at the Pia Fondazione Panico of Tricase, Italy.

To have an imbalanced results and to reduce any bias, a randomization list has been checked.

Probability (p) values will be considered to be statistically significant at the <0.05 level.

There will be recruited 32 patients for Groups. Group 1: Laparoscopic Fascial posterior vaginal duplication with absorbable sutures plus sacral colpopexy mesh placement Vs Group 2: Laparoscopic sacral colpopexy isolated for vaginal posterior prolapse.

All patients will be adequately informed and inserted in the study only after having read and signed an informed consent. Diagnostic, clinical and surgical data of each patient will be prospectively recorded. At the end of the procedure, a schedule will be compiled with intraoperative data. All clinical and histologic data will be recorded prospectively using a database. Pain associated with the procedure will be evaluated by a subjective assessment (analysis of VAS scale values reported by patients at 8 and 24 hours after surgery). Post-operative complications will be evaluated during the first 30 days after surgery according to Dindo's classification.

ELIGIBILITY:
Age ≤ 80 years Patient's informed consent American Society of Anesthesiologists: < class III or IV

No previous major abdominal surgical procedures POP-Q stage > or =III for posterior compartment. No uterine cervix dysplasia or endometrial disorders. No uterine size larger than conform 10 weeks gestation

Max Age: 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
POP-Q | 1 year
  POP-Q evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morciano, Principal Investigator — Pia Fondazione Panico
Locations (1):
- Pia Fondazione Panico, Tricase, Lecce, Italy